CLINICAL TRIAL: NCT02261688
Title: Evaluation of the Influence of Salt Intake on TH17 Interleukin(IL)-17 Producing CD4+ Helper T Cells in Human Subjects
Brief Title: Salt and TH-17 in Healthy Human Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Chief, Cardiovascular Endocrinology Section, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013P002358
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Th17 Helper Immune Cells; Autoimmunity; Salt Intake; Sodium Chloride
MeSH Terms: conditions — Autoimmune Diseases | interventions — Diet, Sodium-Restricted; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects in study (Other): All subjects in study are in a cross-over study with 3 interventions sequentially (low salt diet, low salt diet + IV normal saline, liberal salt diet)
  Interventions: Dietary Supplement: Low salt diet; Dietary Supplement: Low salt diet + IV normal saline; Dietary Supplement: Liberal salt diet

INTERVENTIONS:
Dietary Supplement: Low salt diet — Low salt diet, 10mmoL of sodium per day, for 6 days
Dietary Supplement: Low salt diet + IV normal saline — Low salt diet, 10 mmoL of sodium per day, for 4 days with normal saline infusion x 12 hours per day for 200 mmoL of sodium chloride. Total daily sodium is 210 mmoL/day.
Dietary Supplement: Liberal salt diet — Liberal salt diet targeting 200 mmoL of sodium per day x 7 days

SUMMARY:
The overall goal of this study is to evaluate the association between sodium and TH17 cells in human subjects. The subjects will have levels of TH-17 and various hormones measured on low salt diet, low salt diet with intravenous normal saline, and high salt diet.

DETAILED DESCRIPTION:
In recent years, dietary sodium intake has dramatically increased and has been shown to play an active role in a number of detrimental diseases including hypertension and cardiovascular complications. Additionally, in the developed world, there has been a steady increase in autoimmune diseases. Type 17 helper T cells (Th17) have been shown to play an active role in the development of autoimmune diseases.

Serum glucocorticoid kinase (SGK1) has been shown to influence sodium transport and salt homeostasis in many cell types (Wulf, J. Clin. Invest. 2002; Salker, Nature Med 2011). Prior in vitro and in vivo studies have shown that an increase in salt concentration in the media or dietary salt intake in mice induces SGK1 expression and enhances TH17 cell differentiation and worsens experimental autoimmune encephalomyelitis (EAE), animal model for multiple sclerosis (Kleinewietfeld, Nature 2013; Wu, Nature 2013).

The findings in this study can substantially increase the investigators understanding of environmental factors that modulate the development of autoimmunity in humans. In animal models the worsening effects of a high salt diet on EAE are dramatic. To the investigators knowledge, the proposed study will be the first to determine if salt intake has the same adverse impact in humans. If documented, one could envision the development of a novel treatment approach for human autoimmunity via the regulation of salt intake. Thus, the overall goal of this study is to evaluate the association between sodium and TH17 cells in human subjects. In addition to measuring TH17 cells by flow cytometry the investigators will also measure interleukins such as IL-17a, IL-17f, IL-23 that are important in TH17 differentiation and production.

ELIGIBILITY:
Inclusion Criteria:

* We will seek normal, healthy volunteers age 18-45 years. Participants must be healthy, BMI 18-25.
* We will first recruit male subjects into the pilot study to fully assess the relationship between immune status and salt intake in the absence of hormonal influences (ovulation and menstruation) to establish a baseline understanding before embarking on such a study in women. We will study healthy women subjects in a subsequent later study.

Subjects must have normal laboratory values for:

1. Complete blood count
2. Serum creatinine, sodium, potassium, glucose, liver enzymes
3. Urinalysis
4. Normal ECG

Exclusion Criteria:

We will exclude individuals with:

* Systolic blood pressure > 140 or < 90
* Diastolic blood pressure >90 or < 60
* Creatinine Clearance is abnormal (MDRD formula)
* Known DM, CHF, CAD, PVD, CVA, MI, or RAS.
* Known autoimmune disease (including thyroid disease, asthma, inflammatory bowel disease, rheumatologic diseases)
* Known neurologic disease (i.e. MS)
* Steroid use (oral or inhaled, chronic or within the past 6 months)
* Significant concomitant medical illnesses (cancer, chronic active immunological conditions, etc.)
* If spot Na > 30 after low salt diet
* Current excessive etoh (>10oz/etoh/week)
* Current use of recreational drugs
* Current smokers
* Abnormal labs
* Acute hospitalizations including surgery in the past 6 months
* Chronic use of non-steroidal anti-inflammatory or narcotic medications
* Evidence of ischemia or heart block on screening electrocardiogram (greater than type I-second degree heart block, left bundle branch block, or
* ST-T wave changes in 2 or more contiguous leads)
* Subjects taking any prescription medications (with the exception of birth control pills) or herbal medications will be excluded).
* Ingestion of probiotics within last 3 months
* Antibiotic use within last 3 months
* 1st degree relative with an onset of diabetes or hypertension before the age of 60
* 1st degree relative with autoimmune disease (including thyroid disease, asthma, inflammatory bowel disease, rheumatologic diseases)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
TH-17 levels | 5 days

SECONDARY OUTCOMES:
IL-17 levels | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States